CLINICAL TRIAL: NCT04551157
Title: Early Adjustment Following Open Fracture: the Impact of Viewing Psychoeducational Video Material.
Brief Title: Impact of Psychoeducational Video on Adjustment to Open Fracture.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit during Covid & funding no longer available
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Louise Quarmby, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 263694
Record Dates: First submitted 2020-09-03; First posted 2020-09-16 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Major Trauma
Keywords: major trauma; open fracture; intervention; appearance
MeSH Terms: conditions — Fractures, Open

STUDY DESIGN:
Intervention Model Description: Participants randomised to intervention group (video-viewing) or treatment-as-usual (control) group.
Masking Description: Participants will be made aware at the time of informed consent that they will be randomised to either view the videos or receive treatment-as-usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Viewing (Experimental): Participants will receive the intervention where they will view two patient information videos. The first video will be viewed within the first week of their inpatient stay and the second video will be viewed just before discharge.
  Interventions: Other: Video Viewing
- Treatment as usual (No Intervention): No change to routine care.

INTERVENTIONS:
Other: Video Viewing — Two patient information videos containing practical advice from staff about the recovery process, images of the wound throughout the healing process and ways to cope with the range of emotional responses that patients report following an open fracture.
  Arms: Video Viewing

SUMMARY:
The multi-disciplinary team involved in the care of major trauma patients with open fractures has developed two novel patient information videos. They include practical advice from staff about the recovery process, images of the wound throughout the healing process and ways to cope with the range of emotional responses that patients report following an open fracture. The experiences of previous patients are also included. The aim of this project is to evaluate the impact of viewing these videos on patients' ability to follow treatment recommendations made by the team, as well as their psychological and social functioning, as measured by standardised questionnaire responses. Additionally, the patient's experience of viewing the videos, in terms of how relevant and useful they found them, will be evaluated.

DETAILED DESCRIPTION:
High levels of psychological difficulty are often reported by patients with an open fracture. These patients frequently describe feeling distressed by the initial appearance of their scars and can struggle to adjust and prepare for the challenges they face on discharge from hospital. Patients' expectations about the appearance of their wounds and their role in the recovery process may be aided with access to visual material that the patient and their family can revisit as often as is helpful to them.

Therefore, the multi-disciplinary team involved in the care of these patients has developed two novel patient information videos. They include practical advice from staff about the recovery process, images of the wound throughout the healing process and ways to cope with the range of emotional responses that patients report following an open fracture. The experiences of previous patients are also included. The aim of this project is to evaluate the impact of viewing these videos on patients' ability to follow treatment recommendations made by the team, as well as their psychological and social functioning, as measured by standardised questionnaire responses. Additionally, the patient's experience of viewing the videos, in terms of how relevant and useful they found them, will be evaluated.

All adult patients with an open fracture attending the John Radcliffe Hospital Major Trauma Centre will be eligible to take part (unless they have a diagnosis of dementia, active delirium or traumatic brain injury). Participation will involve completing questionnaires whilst in hospital (within the first week and prior to discharge) and at a routine 3-month follow-up appointment. Patients will be randomly selected to either view the videos or receive treatment as usual. The questionnaire responses of patients in these two groups will be compared to help evaluate the videos.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Fluent in English.
* Diagnosed with an open fracture.
* Inpatient stay of >72 hours.

Exclusion Criteria:

* Participant has a diagnosis of dementia.
* Participant is experiencing delirium.
* Participant has a complete spinal fracture.
* Participant has a traumatic brain injury with a clinically significant presentation.
* Participant is unable to provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes Routine Evaluation 10 (CORE-10) | 3-7 days after hospital admission (Timepoint 1 - baseline)
  The CORE-10 is a brief, generic and easy-to-use measure of psychological distress. It is a self-report questionnaire with ten items about how the respondent has been feeling over the last week, with a 5-point Likert scale (Not at all/Only occasionally/Sometimes/Often/Most of the time). These items cover symptoms (depression, anxiety, trauma, physical problems), functioning (general, social and close relationships sub-domains) and risk to self. All items are summed (items 2 and 3 are reversed scored). The minimum score is 0 and the maximum score is 40, with higher scores indicating higher levels of psychological distress. The clinical cut-off score for general psychological distress is 11.0. The clinical cut-off for depression is 13.0 (sensitivity and specificity values of .92 and 0.72 respectively).
Clinical Outcomes Routine Evaluation 10 (CORE-10) | 7-14 days after admission (Timepoint 2 - prior to discharge)
  The CORE-10 is a brief, generic and easy-to-use measure of psychological distress. It is a self-report questionnaire with ten items about how the respondent has been feeling over the last week, with a 5-point Likert scale (Not at all/Only occasionally/Sometimes/Often/Most of the time). These items cover symptoms (depression, anxiety, trauma, physical problems), functioning (general, social and close relationships sub-domains) and risk to self. All items are summed (items 2 and 3 are reversed scored). The minimum score is 0 and the maximum score is 40, with higher scores indicating higher levels of psychological distress. The clinical cut-off score for general psychological distress is 11.0. The clinical cut-off for depression is 13.0 (sensitivity and specificity values of .92 and 0.72 respectively).
Clinical Outcomes Routine Evaluation 10 (CORE-10) | 3-months post-injury (Timepoint 3 - follow-up)
  The CORE-10 is a brief, generic and easy-to-use measure of psychological distress. It is a self-report questionnaire with ten items about how the respondent has been feeling over the last week, with a 5-point Likert scale (Not at all/Only occasionally/Sometimes/Often/Most of the time). These items cover symptoms (depression, anxiety, trauma, physical problems), functioning (general, social and close relationships sub-domains) and risk to self. All items are summed (items 2 and 3 are reversed scored). The minimum score is 0 and the maximum score is 40, with higher scores indicating higher levels of psychological distress. The clinical cut-off score for general psychological distress is 11.0. The clinical cut-off for depression is 13.0 (sensitivity and specificity values of .92 and 0.72 respectively).
Appearance-Related Psychosocial Distress Scale | 3-7 days after hospital admission (Timepoint 1 - baseline)
  This is an 8-item self-report scale where respondents are asked to disagree or agree to 8 statements about their appearance using a 4-point likert scale (Definitely disagree/Somewhat disagree/Somewhat agree/Definitely agree). The minimum score is 8 and the maximum is 32, which higher scores indicating higher levels of appearance-related psychosocial distress. Klassen and colleagues (2016) used Rasch Measurement Theory (RMT) analysis to assess the psychometric properties of the measure. Person Separation Index (analogous to a reliability index) and Cronbach alpha values were 0.81 and 0.89 respectively. Convergent and predictive validity of this scale have not yet been assessed.
Appearance-Related Psychosocial Distress Scale | 7-14 days after admission (Timepoint 2 - prior to discharge)
  This is an 8-item self-report scale where respondents are asked to disagree or agree to 8 statements about their appearance using a 4-point likert scale (Definitely disagree/Somewhat disagree/Somewhat agree/Definitely agree). The minimum score is 8 and the maximum is 32, which higher scores indicating higher levels of appearance-related psychosocial distress. Klassen and colleagues (2016) used Rasch Measurement Theory (RMT) analysis to assess the psychometric properties of the measure. Person Separation Index (analogous to a reliability index) and Cronbach alpha values were 0.81 and 0.89 respectively. Convergent and predictive validity of this scale have not yet been assessed.
Appearance-Related Psychosocial Distress Scale | 3-months post-injury (Timepoint 3 - follow-up)
  This is an 8-item self-report scale where respondents are asked to disagree or agree to 8 statements about their appearance using a 4-point likert scale (Definitely disagree/Somewhat disagree/Somewhat agree/Definitely agree). The minimum score is 8 and the maximum is 32, which higher scores indicating higher levels of appearance-related psychosocial distress. Klassen and colleagues (2016) used Rasch Measurement Theory (RMT) analysis to assess the psychometric properties of the measure. Person Separation Index (analogous to a reliability index) and Cronbach alpha values were 0.81 and 0.89 respectively. Convergent and predictive validity of this scale have not yet been assessed.
Trauma Screening Questionnaire (TSQ) | 3-7 days after hospital admission (Timepoint 1 - baseline)
  The TSQ is a 10-item self-report questionnaire with items covering the different reactions that sometimes occur after a traumatic event. Respondents are asked to endorse Yes/No to whether or not they have experienced any of the following at least twice in the last week. Predictive validity of respondents who endorsed at least six of the re-experiencing or arousal items (in any combination) was excellent. Sensitivity was 0.86 and specificity was 0.93. Other research by Brewin, Fuchkan, Huntley & Scragg (2010) has indicated low specificity in non-white samples. Specificity was also low if the TSQ was administered early after the trauma but this improved in the eighteen months following the event.
Trauma Screening Questionnaire (TSQ) | 7-14 days after admission (Timepoint 2 - prior to discharge)
  The TSQ is a 10-item self-report questionnaire with items covering the different reactions that sometimes occur after a traumatic event. Respondents are asked to endorse Yes/No to whether or not they have experienced any of the following at least twice in the last week. Predictive validity of respondents who endorsed at least six of the re-experiencing or arousal items (in any combination) was excellent. Sensitivity was 0.86 and specificity was 0.93. Other research by Brewin, Fuchkan, Huntley & Scragg (2010) has indicated low specificity in non-white samples. Specificity was also low if the TSQ was administered early after the trauma but this improved in the eighteen months following the event.
Trauma Screening Questionnaire (TSQ) | 3-months post-injury (Timepoint 3 - follow-up)
  The TSQ is a 10-item self-report questionnaire with items covering the different reactions that sometimes occur after a traumatic event. Respondents are asked to endorse Yes/No to whether or not they have experienced any of the following at least twice in the last week. Predictive validity of respondents who endorsed at least six of the re-experiencing or arousal items (in any combination) was excellent. Sensitivity was 0.86 and specificity was 0.93. Other research by Brewin, Fuchkan, Huntley & Scragg (2010) has indicated low specificity in non-white samples. Specificity was also low if the TSQ was administered early after the trauma but this improved in the eighteen months following the event.
General Adherence Measure | 3-7 days after hospital admission (Timepoint 1 - baseline)
  This is a general measure of patient's adherence to treatment, where respondents are asked how often they were able to adhere to their treatment. It has 5-items and a 6-point Likert response scale (None of the time/A little of the time/Some of the time/A good bit of the time/Most of the time/All of the time). The minimum score is 5 and the maximum score is 24, with higher scores indicating better adherence to treatment. The internal consistency of the measure has been found to be acceptable with a Cronbach's alpha of 0.81 (Hays, n.d).
General Adherence Measure | 7-14 days after admission (Timepoint 2 - prior to discharge)
  This is a general measure of patient's adherence to treatment, where respondents are asked how often they were able to adhere to their treatment. It has 5-items and a 6-point Likert response scale (None of the time/A little of the time/Some of the time/A good bit of the time/Most of the time/All of the time). The minimum score is 5 and the maximum score is 24, with higher scores indicating better adherence to treatment. The internal consistency of the measure has been found to be acceptable with a Cronbach's alpha of 0.81 (Hays, n.d).
General Adherence Measure | 3-months post-injury (Timepoint 3 - follow-up)
  This is a general measure of patient's adherence to treatment, where respondents are asked how often they were able to adhere to their treatment. It has 5-items and a 6-point Likert response scale (None of the time/A little of the time/Some of the time/A good bit of the time/Most of the time/All of the time). The minimum score is 5 and the maximum score is 24, with higher scores indicating better adherence to treatment. The internal consistency of the measure has been found to be acceptable with a Cronbach's alpha of 0.81 (Hays, n.d).
Condition specific statements about treatment and scarring | 3-7 days after hospital admission (Timepoint 1 - baseline)
  This includes 4 statements about the patient's treatment and 10 about their scarring, written by the chief investigator and based on clinical experience. The items address how the patient feels about their treatment, their expectations about ongoing treatment and healing and their role in the recovery process. The items focus on the patient's emotional responses to their scars and their perceptions about the impact the scars may have on their quality of life. These items are on a 4-point agreement scale (Definitely disagree/Somewhat disagree/Somewhat agree/Definitely agree). For the treatment section, the minimum score is 4 and the maximum score is 16, with higher scores indicating better understanding of treatment. and better adjustment/more positive attitudes towards scarring respectively. For the scarring section, the minimum score is 10 and the maximum score is 40, with higher scores indicating better adjustment/more positive attitudes towards scarring respectively.
Condition specific statements about treatment and scarring | 7-14 days after admission (Timepoint 2 - prior to discharge)
  This includes 4 statements about the patient's treatment and 10 about their scarring, written by the chief investigator and based on clinical experience. The items address how the patient feels about their treatment, their expectations about ongoing treatment and healing and their role in the recovery process. The items focus on the patient's emotional responses to their scars and their perceptions about the impact the scars may have on their quality of life. These items are on a 4-point agreement scale (Definitely disagree/Somewhat disagree/Somewhat agree/Definitely agree). For the treatment section, the minimum score is 4 and the maximum score is 16, with higher scores indicating better understanding of treatment. and better adjustment/more positive attitudes towards scarring respectively. For the scarring section, the minimum score is 10 and the maximum score is 40, with higher scores indicating better adjustment/more positive attitudes towards scarring respectively.
Condition specific statements about treatment and scarring | 3-months post-injury (Timepoint 3 - follow-up)
  This includes 4 statements about the patient's treatment and 10 about their scarring, written by the chief investigator and based on clinical experience. The items address how the patient feels about their treatment, their expectations about ongoing treatment and healing and their role in the recovery process. The items focus on the patient's emotional responses to their scars and their perceptions about the impact the scars may have on their quality of life. These items are on a 4-point agreement scale (Definitely disagree/Somewhat disagree/Somewhat agree/Definitely agree). For the treatment section, the minimum score is 4 and the maximum score is 16, with higher scores indicating better understanding of treatment. and better adjustment/more positive attitudes towards scarring respectively. For the scarring section, the minimum score is 10 and the maximum score is 40, with higher scores indicating better adjustment/more positive attitudes towards scarring respectively.

SECONDARY OUTCOMES:
Intervention acceptability and feasibility measure | 7-14 days after admission (Timepoint 2 - prior to discharge)
  This is a 10-item measure developed specifically for the purpose of this study by the chief investigator. Patients are asked to respond to 6 statements on a 4-point agreement scale (Definitively disagree/Somewhat disagree/Somewhat agree/Definitely agree). This includes items such as 'the videos contained information that was relevant to me' and 'I found the videos upsetting to watch'. The minimum score is 6 and the maximum score is 24, with higher scores indicating higher acceptability and feasibility of the intervention. There are an additional 2 items asking the patient whether the time that they viewed video 1 and video 2 respectively was too soon after the injury, about right or too late after the injury.
Intervention acceptability and feasibility measure | 3-months post-injury (Timepoint 3 - follow-up)
  This is a 10-item measure developed specifically for the purpose of this study by the chief investigator. Patients are asked to respond to 6 statements on a 4-point agreement scale (Definitively disagree/Somewhat disagree/Somewhat agree/Definitely agree). This includes items such as 'the videos contained information that was relevant to me' and 'I found the videos upsetting to watch'. The minimum score is 6 and the maximum score is 24, with higher scores indicating higher acceptability and feasibility of the intervention. There are an additional 2 items asking the patient whether the time that they viewed video 1 and video 2 respectively was too soon after the injury, about right or too late after the injury.

CONTACTS AND LOCATIONS:
Overall Officials: May Quarmby, D Clin, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No